CLINICAL TRIAL: NCT06563635
Title: Frequency of Tuberculosis in Psoriasis Patients Using Anti-TNF Therapy During 15 Years of Follow-up.
Brief Title: Frequency of Tuberculosis in Psoriasis Patients
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: E-54022451-050.05.04-116589
Record Dates: First submitted 2023-08-31; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Psoriasis Vulgaris; Tuberculosis
Keywords: psoriasis; tnf inhibitor; tuberculosis
MeSH Terms: conditions — Tuberculosis; Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- etanercept: psoriasis patients receiving etanercept therapy
- infliximab: psoriasis patients receiving infliximab therapy
- adalimumab: psoriasis patients receiving adalimumab therapy

SUMMARY:
Aim of this study is evaluation of patients receiving TNF inhibitor therapy in terms of tuberculosis at the end of 15 years in a single center.

DETAILED DESCRIPTION:
Aim of this study is evaluation of patients receiving TNF inhibitor therapy in terms of tuberculosis at the end of 15 years in a single center. TNF inhibitor therapy may increase the risk for tuberculosis infection. According to medical data in our hospital in last 15 years, tuberculosis rate of psoriasis patients receiving etanercept, adalimumab and infliximab will be compared.

ELIGIBILITY:
Inclusion Criteria:

* psoriasis patients receiving TNF inhibitor therapy

Exclusion Criteria:

* patients without TNF inhibitor therapy

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: psoriasis patients receiving TNF inhibitor therapy in a single center in 15 years
Sampling Method: Non-Probability Sample
Enrollment: 719 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
tuberculosis rate | patients from June 2007 to January 2023, up to 15 years
  number of patients with tuberculosis infection after receiving TNF inhibitor therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University Hospital, Istanbul, Turkey (Türkiye)